CLINICAL TRIAL: NCT01799421
Title: Predictive Models of Risk Assessment of Febrile Neutropenia and Grade 3-4 Neutropenia in Patients With Non-hematological Cancer Treated With Conventional Chemotherapy.
Brief Title: Risk Assessment of Febrile Neutropenia and Grade 3-4 Neutropenia in Patients With Non-hematological Cancer Treated With Conventional Chemotherapy
Acronym: NEURISK
Status: Completed | Type: Observational
Sponsor: Asociación para el Fomento de la Investigación y el Desarrollo Integral de la Oncología (Other)
Responsible Party: Sponsor
Other Study IDs: NEURISK
Record Dates: First submitted 2013-02-23; First posted 2013-02-26 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Non-hematologic Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-haematologic cancer

SUMMARY:
The purpose of this study is to identify prognostic factors and to develop predictive models of risk of febrile neutropenia and neutropenia grade 3/4 in patients with solid tumors receiving chemotherapy with schemas that have an inherent risk of febrile neutropenia of 10-20%.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years
* Histologically confirmed solid tumor.
* Subjects who have not received chemotherapy and / or radiotherapy in the last 3 months.
* Subject to initiate a chemotherapy (ie, cycle 1, day 1)
* The chemotherapy regimen should have an inherent risk of febrile neutropenia of 10-20%.
* Planning a minimum of 3 cycles chemotherapy.
* Adequate bone marrow reserve defined by: leukocytes ≥ 3,000 / mm3, platelets ≥ 100.000/mm3; neutrophils ≥ 1,500 / mm3.
* Adequate hepatic and renal function, defined by: bilirubin <1.5 times the normal value, ALT and AST <3 times the normal range (both can be elevated up to 5 times the normal value in patients with known liver metastases); creatinine <1.5 times upper normal value
* ECOG ≤ 2.
* Informed consent

Exclusion Criteria:

* Patients under treatment with an investigational treatment.
* Active infection in the last 72 h before starting chemotherapy.
* Indication of chemotherapy dose intensity or chemotherapy included in the risk rating of febrile neutropenia <10% or >20%.
* Patients with concomitant chemoradiotherapy.
* Patients being treated with biological drugs in monotherapy.
* Any other condition causing neutropenia.
* History of bone marrow transplant or stem cells.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-hematologic cancer that will start chemotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Identify predictive models about the risk of febrile neutropenia and neutropenia grade 3/4 in patients with non-hematologic cancer | 6 months

SECONDARY OUTCOMES:
Occurrence of serious adverse events | 6 months
Analyze costs to treat febrile neutropenia and neutropenia grade 3/4 | 6 months
Analyze the risk of mortality due to febrile neutropenia and neutropenia grade 3/4 during the chemotherapy treatment | 6 months
  A Cox proportional hazards regression will be used to evaluate the risk of mortality due to febrile neutropenia and neutropenia grade 3/4 during chemotherapy treatment.
Evaluate impact of febrile neutropenia and neutropenia grade 3/4 in treatment compliance | 6 months
  The impact of febrile neutropenia and neutropenia grade 3/4 in treatment compliance (yes/no) will be evaluated using a chi-square test.

CONTACTS AND LOCATIONS:
Locations (20):
- Spain (20):
  - Hospital Teresa Herrera, A Coruña, A coruña
  - Hospital Universitario Albacete, Albacete, Albacete
  - Hospital Clínico Universitario San Juan de Alicante, Alicante, Alicante
  - Hospital Quirón, Barcelona, Barcelona
  - Hospital de Basurto, Basurto, Bilbao
  - Hospital San Pedro de Alcántara, Cáceres, Cáceres
  - Hospital de Jerez, Jerez de la Frontera, Cádiz
  - Hospital Dr. Josep Trueta, Girona, Girona
  - Hospital Virgen de las Nieves, Granada, Granada
  - Hospital de Donosti, San Sebastián, Guipuzcua
  - Hospital de Lugo, Lugo, Lugo
  - Hospital Morales Meseger, Murcia, Murcia
  - Hospital de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Ourense, Ourense, Ourense
  - Hospital Xeral, Vigo, Pontevedra
  - Hospital de Santa Tecla, Tarragona, Tarragona
  - Hospital Virgen de la Salud, Toledo, Toledo
  - Hospital Arnau de Vilanova, Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia, Valencia
  - Hospital Clínico de Valladolid, Valladolid, Valladolid